CLINICAL TRIAL: NCT04808609
Title: A Pilot Trial of a Smoking Cessation App in People Living With HIV (PLWH)
Brief Title: Smoking Cessation Pilot for People Living With HIV (PLWH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Professor of Disease Prevention and Health Promotion (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAS6990
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation; Smoking; Smoking Behaviors; Smoking Reduction; Smoking, Tobacco; Smoking, Cigarette; Hiv; HIV/AIDS
Keywords: Smoking; Smoking Cessation; Smoking Behaviors; Smoking Reduction; Tobacco; Cigarette; PLWH; HIV; HIV/AIDS; mHealth; Mobile Health; Lumme; Pilot
MeSH Terms: conditions — Smoking Cessation; Smoking; Smoking Reduction; Tobacco Smoking; Cigarette Smoking; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): The Intervention group receives standard smoking cessation counseling and nicotine replacement therapy AND access to the Lumme app that tracks smoking behaviors and provides cessation support.
  Interventions: Device: Lumme mobile phone application; Behavioral: Standard of Care
- Control (Other): The Control group receives standard smoking cessation counseling and nicotine replacement therapy
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Device: Lumme mobile phone application — Lumme mobile phone app provides smoking cessation support and tracks smoking behaviors
  Arms: Intervention
Behavioral: Standard of Care — Smoking cessation counseling and nicotine replacement therapy

SUMMARY:
The overall goal of this pilot study is to evaluate the feasibility of the Lumme smartphone app for smoking cessation in people living with HIV (PLWH) and evaluate its effect on smoking cessation. Mobile health (mHealth) technology can be used for achieving health equity in vulnerable groups because it is a widely available and relatively inexpensive tool for health behavior change and can be adapted to meet the needs of its end-users. Therefore, a mHealth intervention such as the Lumme App proposed through this study is timely, relevant, scalable and likely to improve health outcomes in PLWH who smoke.

DETAILED DESCRIPTION:
Of the approximately one million persons living with HIV (PLWH) in the United States (U.S.), it is estimated that between 34-47% smoke cigarettes, around three times the prevalence (12.5%) observed in the general U.S. adult population. Consequently, PLWH experience substantial tobacco-related morbidity and mortality. In PLWH, after achieving and maintaining a suppressed viral load, smoking cessation is the next most important health behavior to maximize both quality of life and life expectancy. Given the high prevalence of cigarette smoking among PLWH and the benefit of smoking cessation, there is an urgent need for swift action to intervene to reduce tobacco use rates. However, evidence to improve tobacco cessation among PLWH is inadequate. Given the need for improving smoking cessation in PLWH, and the great promise of mHealth tools, this research study will assess smoking behaviors in people living with HIV and the subsequent efficacy of mHealth intervention for improving tobacco cessation.

ELIGIBILITY:
Inclusion Criteria:

* PLWH
* ≥ 18 years old
* own an Android smartphone
* understand and read English
* not pregnant or breastfeeding
* permanent contact information
* smokes greater than or equal to 5 cigarettes per day for the past 30 days
* interested in quitting smoking within 30 days
* blow ≥ 6 carbon monoxide (CO) into a breath analyzer at baseline

Exclusion Criteria:

* self-report being HIV-negative or unknown status
* pregnant, breastfeeding, or planning to become pregnant during the study period
* planning to move within 3 months of enrollment
* a positive history of a medical condition that precludes use of the nicotine patch
* current use of nicotine replacement therapy or other smoking cessation medications
* current enrollment in another smoking cessation program
* blows ≤ 5 CO into a breath analyzer at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, RN, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Schnall R, Liu J, Alvarez G, Porras T, Ganzhorn S, Boerner S, Huang MC, Trujillo P, Cioe P. A Smoking Cessation Mobile App for Persons Living With HIV: Preliminary Efficacy and Feasibility Study. JMIR Form Res. 2022 Aug 18;6(8):e28626. doi: 10.2196/28626. PMID 35980739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an existing database of persons living with HIV who had participated in earlier studies and agreed to be re-contacted for future studies and posting flyers at a local HIV clinic between 9/29/2020 and 4/19/2021. The first participant was enrolled 10/6/2020 and the final participant was enrolled 4/19/2021.
Pre-assignment Details: All 40 enrolled participants were randomized.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 20 | 20
Completed | 20 | 17
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Administrative Withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.2) | 54.0 (8.5) | 53.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 13 | 18 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 18 | 31
  White | 0 | 1 | 1
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Exhaled Carbon Monoxide in parts per million [Mean (Standard Deviation); unit: parts per million] — Participants provided a breath sample at baseline to assess exhaled carbon monoxide in parts per million
  parts per million | 14.5 (6.5) | 13.1 (6.3) | 13.8 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biochemically Verified 7-day Point Prevalence Smoking/Tobacco Abstinence
Description: 7-day point prevalence abstinence was calculated as the percentage of participants who reported no smoking/tobacco use in the 7 days prior to their 12-week follow-up visit biochemically verified by exhaled Carbon Monoxide (eCO) collected at 12 weeks. Participants with eCO levels <6 parts per million (ppm) at 12 weeks were classified as abstinent while participants with eCO levels ≥6ppm at 12 weeks were classified as not abstinent.
Time Frame: Baseline, 12 weeks follow up
Population: All participants who provided follow up data at 12 weeks were included in the outcome analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 17
percentage of participants | 15.0 [3.2 to 37.9] | 11.8 [1.5 to 36.4]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — feasibility test; p = 0.77, Fisher Exact; Risk Ratio (RR) = 1.27, 95% CI 2-sided [0.24 to 6.76], Standard Error of Mean 1.63

2. Secondary Outcome: Percentage of Participants With Self-reported 7-day Point Prevalence Abstinence at 12 Weeks
Description: 7-day point prevalence abstinence was calculated as the percentage of participants who reported no smoking/tobacco use in the 7 days prior to their 12-week follow-up visit.
Time Frame: Baseline, 12 weeks follow up
Population: All participants who provided follow up data at 12 weeks were included in the outcome analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 17
percentage of participants | 30.0 [11.9 to 54.3] | 23.5 [6.8 to 49.9]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — feasibility test; p = 0.66, Chi-squared; Risk Ratio (RR) = 1.27, 95% CI 2-sided [0.43 to 3.78], Standard Error of Mean 0.84

3. Secondary Outcome: Change in eCO in Ppm From Baseline to 12-week Follow-up
Description: Exhaled Carbon Monoxide (eCO) was measured via Micro +TM basic Smokerlyzer® in parts per million (ppm) and collected at Baseline and at 12-week Follow-up. Theoretically possible result values range from 0 to 150 ppm with higher values indicating more eCO. Mean change for this study was calculated as Baseline eCO value minus 12-week Follow-up eCO value such that positive mean values indicate a decrease in eCO from Baseline to 12-week Follow-up.
Time Frame: Baseline to 12-week Follow-up
Population: All participants who provided follow up data at 12 weeks were included in the outcome analysis
Measure: Mean (95% Confidence Interval); unit: parts per million (ppm)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 17
parts per million (ppm) | 3.35 [-0.22 to 6.92] | 2.12 [-0.9 to 5.14]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — feasibility test; p = 0.59, t-test, 2 sided; Cohen's D = 0.21, 95% CI 2-sided [-0.44 to 0.86], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Intervention vs Control; Results from Paired T-Test assessing the with-subject time effect on exhaled CO in ppm from baseline to 12 weeks; Test type: Other — feasibility; p = 0.02, t-test, 1 sided; Cohen's D = 0.41, 95% CI 2-sided [0.07 to 0.74], Standard Error of Mean 0.17

4. Secondary Outcome: Change in Center for Epidemiologic Studies Depression Scale (CES-D) Score
Description: The CES-D measure contains 20 items asking respondents to rate how often over the past week they experienced depression-associated symptoms. Response options are coded as: 0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time. Scores are calculated by reversing scores for positive statements and adding all responses together. Scores range from 0 to 60, with higher scores indicating greater presence of depressive symptoms.
Time Frame: Baseline, 12-week Follow-up
Population: All participants who provided follow up data at 12 weeks were included in the outcome analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 17
score on a scale | 16.6 [10.8 to 22.3] | 14.8 [10.8 to 18.7]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — feasibility test; p = 0.61, t-test, 2 sided; Cohen's D = 0.16, 95% CI 2-sided [-0.46 to 0.78], Standard Error of Mean 0.31

5. Secondary Outcome: Self-reported Number of Cigarettes Smoked Daily at Baseline
Description: During baseline visit, participants were asked to report how many cigarettes they smoked daily during the past 30 days.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: cigarettes smoked per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
cigarettes smoked per day | 11.9 [9.5 to 14.3] | 11.0 [9.3 to 12.7]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — feasibility test; p = 0.55, t-test, 2 sided; Cohen's D = 0.19, 95% CI 2-sided [-0.42 to 0.80], Standard Error of Mean 0.31

6. Secondary Outcome: CAGE Substance Abuse Screening Tool Score at Baseline
Description: The CAGE Substance Abuse Screening Tool contains 4 questions with binary answer options: 1 = Yes, 0 = No. Scores are calculated by adding response values. Scores range from 0 to 4 with higher scores indicating alcohol problems. CAGE stands for the 4 question names: Cut down, Annoyed, Guilty, and Eye-opener
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
score on a scale | 0.9 [0.2 to 1.6] | 0.9 [0.3 to 1.5]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — feasibility test; p = 0.99, t-test, 2 sided; Cohen's D = 0.004, 95% CI 2-sided [-0.61 to 0.62], Standard Error of Mean 0.31

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the entire study period, an average of 3 months from baseline visit to follow-up visit.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04808609/Prot_SAP_000.pdf